CLINICAL TRIAL: NCT01159106
Title: The Use of NAVA vs. Pressure Support During Asynchrony in Children
Brief Title: The Use of Neurally Adjusted Ventilatory Assist (NAVA) Versus Pressure Support During Asynchrony in Children
Acronym: NAVAChildren
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Pedro de la Oliva, Hospital Universitario La Paz
Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: HULP-PI-3132
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2010-07-09 (Estimated); Status verified 2010-07

CONDITIONS: Patient/Ventilator Asynchrony
Keywords: Positive Pressure Ventilation; Neurally Adjusted Ventilatory Assist; Patient/ventilator Asynchrony; Pediatric patient; Infant
MeSH Terms: conditions — Patient-Ventilator Asynchrony | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Pressure Support Ventilation — Spontaneous mode of ventilation whereby the patient initiates the breath and the ventilator delivers support with the preset pressure value
Other: Neurally adjusted ventilatory assist (NAVA) — Gas delivery from the mechanical ventilator is triggered, controlled and cycled by the diaphragmatic EMG signal (Edi).
  The ventilator is aware of the change in diaphragmatic EMG by the insertion of a specially designed nasogastric tube with EMG electrodes that cross the diaphragm.

SUMMARY:
The aim of the current study is to compare the application neurally adjusted ventilatory assist (NAVA) to optimize pressure support ventilation in 12 pediatric patients.

DETAILED DESCRIPTION:
Asynchrony during assisted ventilation in children is common because of the presence of uncuffed artificial airways and their rapid ventilatory rate with small volumes compared to adults.As a result, the most common approach to ventilatory support in children is pressure ventilation, since pressure targeted ventilation allows gas delivery to vary based on patient demand. In addition, many manufacturers have incorporated adjuncts designed to improve synchrony in pressure targeted ventilation. Most of today's ICU ventilators incorporate rise time and control of the breath termination criteria in pressure ventilation by either altering inspiratory time directly or adjusting the inspiratory flow termination criteria in pressure support ventilation. In addition, careful adjustment of trigger sensitivity, and insuring driving pressure is appropriately set to avoid large tidal volumes improves synchrony in many patients. However, in spite of all of these potential adjustments many pediatric patients are still asynchronous.

A recently released new mode of ventilation, NAVA (neurally adjusted ventilatory assist) is designed to reduce the asynchrony that exists between the ventilator and the patient. With NAVA, gas delivery from the mechanical ventilator is triggered, controlled and cycled by the diaphragmatic EMG signal (Edi). The ventilator is aware of the change in diaphragmatic EMG by the insertion of a specially designed nasogastric tube (NGT) with EMG electrodes that cross the diaphragm. This NGT also functions similar to any standard NGT. NAVA is used to control all aspects of assisted ventilatory support. A number of preliminary studies in neonates and pediatric patients have demonstrated that patient ventilator synchrony is improved with the application of NAVA. In general, tidal volumes delivered by the ventilator are decreased, respiratory rates increased and peak inspiratory pressures decreased. In these studies, triggering and cycling of the ventilator are controlled by the diaphragmatic EMG in more than 70 % of the time. If the EMG signal does not activate or terminate positive pressure backup flow/pressure/time signal, control gas delivery -as is customary in standard modes of ventilatory support- takes over.

We hypothesize that the use of NAVA will improve trigger and flow synchrony in children and insure that tidal volumes are normalized (6 to 8 ml/kg) in these patients.

Asynchrony will be studied in 12 mechanically ventilated pediatric patients in the Pediatric ICU at Hospital Universitario Materno-Infantil La Paz in Madrid, Spain.

The study protocol has 5 phases

* Phase 0: patient asynchrony documentation and 10 min recording
* Phase 1: NAVA catheter insertion and 10 min recording in basal ventilatory mode after 20 min stabilization
* Phase 2: Pressure support is optimized and 10 min recording after 20 min stabilization
* Phase 3: NAVA mode ventilation and 10 min recording after 20 min stabilization
* Phase 4: Pressure support ventilation and 10 min recording after 20 min stabilization

ELIGIBILITY:
Inclusion Criteria:

* Trigger asynchrony
* Breath initiation asynchrony
* Breath termination asynchrony
* Patient ventilated by Servo i (Maquet Critical Care AB,Solna,Sweden)
* Patients breathing spontaneously with no control breaths

Exclusion Criteria:

* Shock
* Agitation
* Asynchrony caused by pain
* Abundant tracheal secretions

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Level of asynchrony | 3 hours
  Number of each defined forms of asynchrony per minute during pressure support and during NAVA Six forms of asynchrony will be identified during optimal pressure support and optimal NAVA: trigger asynchrony, breath initiation asynchrony and breath termination asynchrony, demand asynchrony, inspiratory asynchrony and neuro-asynchrony

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Kacmarek, PhD RRT FCCM, Study Director — Massachusetts General Hospital; Pedro de la Oliva, MD PhD, Principal Investigator — Hospital Universitario La Paz; Jesus Villar, MD PhD, Principal Investigator — Hospital Universitario Dr. Negrin; Demet Suleymanci, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

REFERENCES:
- [Background] Beck J, Tucci M, Emeriaud G, Lacroix J, Sinderby C. Prolonged neural expiratory time induced by mechanical ventilation in infants. Pediatr Res. 2004 May;55(5):747-54. doi: 10.1203/01.PDR.0000119368.21770.33. Epub 2004 Jan 22. PMID 14739354
- [Background] Spahija J, de Marchie M, Albert M, Bellemare P, Delisle S, Beck J, Sinderby C. Patient-ventilator interaction during pressure support ventilation and neurally adjusted ventilatory assist. Crit Care Med. 2010 Feb;38(2):518-26. doi: 10.1097/CCM.0b013e3181cb0d7b. PMID 20083921
- [Background] Breatnach C, Conlon NP, Stack M, Healy M, O'Hare BP. A prospective crossover comparison of neurally adjusted ventilatory assist and pressure-support ventilation in a pediatric and neonatal intensive care unit population. Pediatr Crit Care Med. 2010 Jan;11(1):7-11. doi: 10.1097/PCC.0b013e3181b0630f. PMID 19593246
- [Derived] de la Oliva P, Schuffelmann C, Gomez-Zamora A, Villar J, Kacmarek RM. Asynchrony, neural drive, ventilatory variability and COMFORT: NAVA versus pressure support in pediatric patients. A non-randomized cross-over trial. Intensive Care Med. 2012 May;38(5):838-46. doi: 10.1007/s00134-012-2535-y. Epub 2012 Apr 6. PMID 22481227